CLINICAL TRIAL: NCT06460935
Title: The Effect of Online Sexual Health Training Given to Nursing Students With the PLISSIT Model on Knowledge, Attitude and Self-Efficacy
Brief Title: The Effect of Online Sexual Health Training Given to Nursing Students on Knowledge, Attitude and Self-Efficacy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, CEYDA SU GUNDUZ, Research Assistant, Marmara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 26.10.2023/101
Record Dates: First submitted 2024-06-11; First posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Nursing Education; Nursing Students; Randomized Controlled Trial; Sexual Health
Keywords: Distance learning; Nursing education; Nursing students; Randomized controlled trial; Sexual health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: PLISSIT Group (Experimental): Nursing students in this group will be given online sexual health training. The training will last for 5 weeks. The training is 20 hours in total. During the training, students will learn the PLISSIT model and evaluate cases involving using this model. Questionnaire will be applied before the training after the training
  Interventions: Behavioral: sexual health training
- No Intervention: Control group (No Intervention): Nursing students in this group will not be subjected to any application and will continue their routine nursing lessons. The questionnaire will be administered to the control group before the training given to the experimental group after the training.

INTERVENTIONS:
Behavioral: sexual health training — The 20-hour sexual health training will be given online for 5 weeks. Case discussions using the Plissit Model will be held in the training content.
  Arms: Experimental: PLISSIT Group

SUMMARY:
Nurses play an important role in providing sexual health care to individuals. In this study, online sexual health training will be implemented in an innovative way by supporting the use of models in the process of providing sexual counseling to the patients of nursing students. The most commonly used PLISSIT model will be taught to nursing students while providing sexual counseling to patients and its effectiveness will be determined.

DETAILED DESCRIPTION:
Nurses play an important role in providing sexual health care to individuals. In this study, online sexual health training will be implemented in an innovative way by supporting the use of models in the process of providing sexual counseling to the patients of nursing students. The most commonly used PLISSIT model will be taught to nursing students while providing sexual counseling to patients and its effectiveness will be determined. The research is planned to be pre-test post-test comparative, randomized, with one experiment and one control group, ın order to determine the effect of online sexual health training given to nursing students with the PLISSIT model on the myths about sexuality, sexual health care knowledge, sexual health care attitude and sexual health care self-efficacy. This research will be carried out between November 2023 and December 2023 with the participation of fourth grade students studying at Marmara University Faculty of Health Sciences, Department of Nursing. Students who is suitable the inclusion criteria will be randomized to the experimental (n=30) and control groups (n=30). The data of the research will be obtained by using "Student Information Form", Sexual Health Care Questionnaire, which includes 3 scales as "Sexual Health Care Knowledge Scale", "Sexual Health Care Attitude Scale", "Sexual Health Care Self-Efficacy Scale" and "Sexual Myths Scale" and "Student Opinion Form on Sexual Health Education". Ethical permission and institutional permission were obtained.During the research, while the control group receives routine training, the experimental group will be given online sexual health training including 20 hours of PLISSIT model teaching by the researcher. The data of the research will be obtained by using the data collection form before the training, after the training.

ELIGIBILITY:
Inclusion Criteria:

* Being a senior nursing student,
* Having sufficient Turkish speaking and understanding skills,
* Agreeing to participate in sexuality education on the online platform,
* Sufficient or unlimited internet access,
* Having any computer, tablet or smart phone,
* Being willing to participate in the research

Exclusion Criteria:

* Desire to leave the research,
* Incomplete filling of data collection forms,
* Not attending the training given in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2023-11-04 (Actual); Primary Completion 2023-11-04 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Knowledge of Sexual Healthcare Scale | baseline, week 8
  The scale was designed to measure the knowledge of nursing students about sexual health care. The scale consists of 31 items. Each item was rated as "yes", "no" and "I don't know". 1 point is given for the correct answer, 0 points for the wrong answer and the answer I don't know. A score between 0-31 can be obtained from the scale.
Self Efficacy for Sexual Healthcare Scale | baseline, week 8
  The scale measures nursing students' self-efficacy in providing sexual health services. The scale consists of 3 sub dimensions and a total of 15 items. Each item is rated on a 5-point Likert scale ranging from 1= strongly disagree, 2= disagree, 3= undecided, 4= agree, 5= strongly agree. The total score ranges from 15 to 75 points.
Attitude to Sexual Healthcare Scale | baseline, week 8
  The scale determines the attitudes of nursing students towards sexual health services. The scale consists of 3 subdimensions and a total of 18 questions. Each item on the 5-point Likert scale is rated as 5 = strongly agree, 4 = agree, 3 = undecided, 2 = disagree, and 1 = strongly disagree. The scores that can be obtained from the scale vary between 18 and 90.

SECONDARY OUTCOMES:
Student Opinion Form on Sexual Health Education | baseline, week 8
  It determines the thoughts of the students about the model taught in education and the satisfaction of the students from the education.
Sexual Myths Scale | baseline, week 8
  The scale has been reported to be a useful tool to reveal whether a person's knowledge is based on sexual myths. In this 5-point Likert-type scale, consisting of 28 items, statements are evaluated between "1 points (I never agree), "5 points (I totally agree). The scale consists of 8 sub-dimensions and 28 items. The total score that can be obtained from the scale can vary between 28-140.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No